CLINICAL TRIAL: NCT05232344
Title: Sexual Intercourse and Vaginal Absorption of Progesterone : Cross-over Prospective Study
Brief Title: Sexual Intercourse and Vaginal Absorption of Progesterone
Acronym: SexVAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: IBSA Institut Biochimique SA (Industry); Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RECHMPL21_0182; 2021-A01552-39 (Other: n° ID-RCB)
Record Dates: First submitted 2022-01-14; First posted 2022-02-09 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Infertility
Keywords: Progesterone; Vaginal absoption; Intercourse; Assisted reproductive technology
MeSH Terms: conditions — Infertility; Coitus | interventions — Estradiol; Progesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Estradiol / Progesterone treatment (Experimental): Estradiol (Provames®, 3 mg morning and evening, or 6 mg per day) Vaginal progesterone (400 mg, Progestan®, evening and morning, ie 800 mg per day).
  Interventions: Drug: Estradiol / Progesterone; Behavioral: Sexual event

INTERVENTIONS:
Drug: Estradiol / Progesterone — Treatment with estradiol (Provames®, 3 mg morning and evening, or 6 mg per day) will start on the 1st or 2nd day of her period. This treatment is continued until the end of the study (discontinuation treatment after the blood test taken on Day 7). After ten days of minimum estradiol treatment (and up to 7 days later to be working days), vaginal progesterone treatment will start in the evening on Day 0 (400 mg, Progestan®, evening and morning, ie 800 mg per day).
Behavioral: Sexual event — A sexual intercourse (protected or not protected by condoms) will take place in a pre-defined order for each participant within one hour of the administration of the progesterone ovum on the evening of Day 2 and Day 6.

SUMMARY:
The objective of this project is to compare the vaginal absorption of progesterone administered in the vaginal ovum by measuring progesteroneemia in 3 situations (or "sexual event"): abstinence, sex protected by condoms and unprotected sex.

DETAILED DESCRIPTION:
Progesterone plays a key role in embryo implantation and maintenance of pregnancy.

In the context of Assisted Reproduction (ART), support for the luteal phase is often necessary and readily provided by the administration of progesterone, mainly vaginal in Europe.

Optimal absorption is essential because low progesterone levels are associated with the chances of lowered pregnancies.

However, it has been shown that vaginal absorption can be reduced following unprotected sex.

Would the use of a condom prevent this alteration of vaginal absorption?

ELIGIBILITY:
Inclusion Criteria:

* Couples, volunteers, on an AMP journey
* Having sexual intercourse with a low risk of transmission of sexually transmitted infection
* Free and informed consent to participate in the study

Inclusion criteria specific to women:

* aged 18 to 40 inclusive

Exclusion Criteria:

Exclusion criteria specific to women:

* Currently taking hormone therapy that may alter progesteroneemia
* Pathology that can modify progesteroneemia
* Body mass index greater than or equal to 32 kg / m2
* Contraindication to the use of hormone replacement therapy
* Known intolerance to vaginal progesterone
* Pregnant woman (βHCG assay positive) or breastfeeding

Exclusion criteria specific to men:

* Erectile or ejaculatory disorder

Exclusion criteria specific to couples:

* Person with poor oral and/or written French comprehension
* Person who for psychological, social, family or geographical reasons could not be followed regularly
* Vulnerable person (Article L1121-6 of the Public Health Code)
* Protected person or unable to give consent
* Person involvment in another clinical research
* Person not affiliated with a French social security scheme or beneficiary of such a scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-04-13 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Progesterone dosage 1 | Change from Baseline progesterone (Day 2) at Day 3
  Change from baseline plasma progesterone (day 2), 11 hours after administration of progesterone vaginal capsules (400 mg) and protected or unprotected intercourse within one hour of progesterone administration, at day 3
Progesterone dosage 2 | Change from Baseline progesterone (Day 2) at Day 7
  Change from baseline plasma progesterone (day 2), 11 hours after administration of progesterone vaginal capsules (400 mg) and protected or unprotected intercourse within one hour of progesterone administration, at day 7

CONTACTS AND LOCATIONS:
Overall Officials: Noémie RANISAVJLEVIC, MD, Study Director — CHU de Montpellier
Locations (1):
- CHU de Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alsbjerg B, Thomsen L, Elbaek HO, Laursen R, Povlsen BB, Haahr T, Humaidan P. Progesterone levels on pregnancy test day after hormone replacement therapy-cryopreserved embryo transfer cycles and related reproductive outcomes. Reprod Biomed Online. 2018 Nov;37(5):641-647. doi: 10.1016/j.rbmo.2018.08.022. Epub 2018 Oct 6. PMID 30385142
- [Background] Cicinelli E, de Ziegler D, Bulletti C, Matteo MG, Schonauer LM, Galantino P. Direct transport of progesterone from vagina to uterus. Obstet Gynecol. 2000 Mar;95(3):403-6. doi: 10.1016/s0029-7844(99)00542-6. PMID 10711552
- [Background] Cedrin-Durnerin I, Isnard T, Mahdjoub S, Sonigo C, Seroka A, Comtet M, Herbemont C, Sifer C, Grynberg M. Serum progesterone concentration and live birth rate in frozen-thawed embryo transfers with hormonally prepared endometrium. Reprod Biomed Online. 2019 Mar;38(3):472-480. doi: 10.1016/j.rbmo.2018.11.026. Epub 2019 Jan 5. PMID 30642638
- [Background] Gaggiotti-Marre S, Martinez F, Coll L, Garcia S, Alvarez M, Parriego M, Barri PN, Polyzos N, Coroleu B. Low serum progesterone the day prior to frozen embryo transfer of euploid embryos is associated with significant reduction in live birth rates. Gynecol Endocrinol. 2019 May;35(5):439-442. doi: 10.1080/09513590.2018.1534952. Epub 2018 Dec 26. PMID 30585507
- [Background] Hussain A, Ahsan F. The vagina as a route for systemic drug delivery. J Control Release. 2005 Mar 21;103(2):301-13. doi: 10.1016/j.jconrel.2004.11.034. Epub 2005 Jan 13. PMID 15763615
- [Background] Labarta E, Mariani G, Holtmann N, Celada P, Remohi J, Bosch E. Low serum progesterone on the day of embryo transfer is associated with a diminished ongoing pregnancy rate in oocyte donation cycles after artificial endometrial preparation: a prospective study. Hum Reprod. 2017 Dec 1;32(12):2437-2442. doi: 10.1093/humrep/dex316. PMID 29040638
- [Background] Merriam KS, Leake KA, Elliot M, Matthews ML, Usadi RS, Hurst BS. Sexual absorption of vaginal progesterone: a randomized control trial. Int J Endocrinol. 2015;2015:685281. doi: 10.1155/2015/685281. Epub 2015 Feb 3. PMID 25713585
- [Background] Sator M, Radicioni M, Cometti B, Loprete L, Leuratti C, Schmidl D, Garhofer G. Pharmacokinetics and safety profile of a novel progesterone aqueous formulation administered by the s.c. route. Gynecol Endocrinol. 2013 Mar;29(3):205-8. doi: 10.3109/09513590.2012.736560. Epub 2012 Nov 6. PMID 23127204
- [Background] van der Linden M, Buckingham K, Farquhar C, Kremer JA, Metwally M. Luteal phase support for assisted reproduction cycles. Cochrane Database Syst Rev. 2015 Jul 7;2015(7):CD009154. doi: 10.1002/14651858.CD009154.pub3. PMID 26148507
- [Background] Yovich JL, Conceicao JL, Stanger JD, Hinchliffe PM, Keane KN. Mid-luteal serum progesterone concentrations govern implantation rates for cryopreserved embryo transfers conducted under hormone replacement. Reprod Biomed Online. 2015 Aug;31(2):180-91. doi: 10.1016/j.rbmo.2015.05.005. Epub 2015 May 18. PMID 26099447